CLINICAL TRIAL: NCT03167515
Title: A Multicenter Study of 074-6751 Lotion in Subjects With Moderate Plaque Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ferndale Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 074-6751-001
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- 074-6751 Lotion (Experimental)
  Interventions: Device: 074-6751 Lotion

INTERVENTIONS:
Device: 074-6751 Lotion — Apply lotion once in the morning and once in the evening daily at approximately the same time every day with 12 hours between doses. Apply the lotion only to the active psoriatic lesions, as instructed by your study doctor.

SUMMARY:
The primary objective of this study is to determine the efficacy and safety of 074-6751 Lotion applied twice daily for four weeks (28 days) in clinical subjects with moderate plaque psoriasis.

DETAILED DESCRIPTION:
Skin diseases that cause swelling like psoriasis can be improved by using products applied to cover the skin, keeping the skin moist. Keeping the skin moist will ease the local signs and symptoms, such as skin redness, scaling, and itching in patients with plaque psoriasis. Researchers are testing 074-6751 Lotion in clinical subjects with moderate plaque psoriasis to see if it can act as a protective barrier for the skin so the skin remains moist and heals over time.

074-6751 Lotion is an investigational device. Eligible clinical subjects will be enrolled in the study and apply 074-6751 Lotion twice daily to all psoriasis plaques in the assigned Treatment Area for 28 days. Efficacy will be assessed in the Treatment Area by Investigator's Global Association (IGA) score, clinical signs of psoriasis, pruritus, and percent BSA affected. Safety will be assessed by adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or non-pregnant female and at least 18 years of age.
2. Subject has provided written informed consent.
3. Females must be post-menopausal, surgically sterile, or using an effective method of birth control.
4. Subject has a clinical diagnosis of stable plaque psoriasis.
5. Subject is willing and able to apply the test article as directed, comply with study instructions and commit to all follow-up visits for the duration of the study.
6. Subject, in the investigator's opinion, is in good general health and free of any disease state, skin condition, or physical condition that might impair evaluation of psoriasis, would require use of interfering therapy (e.g., topical, systemic, or surgical).

Exclusion Criteria:

1. Subject is pregnant, lactating, or is planning to become pregnant during the study.
2. Subject has spontaneously improving or rapidly deteriorating plaque psoriasis.
3. Subject has guttate, pustular, erythrodermic, or other non-plaque forms of psoriasis.
4. Subject has used any of the following topical preparations or procedures in the

   Treatment Area:
   * Emollients/moisturizers within four days prior to Visit I;
   * Topical anti-psoriatic drugs on the body (excluding the scalp) within 14 days of Visit 1; or
   * Phototherapy ( including laser), photo-chemotherapy or other forms of photo based therapy for the treatment of their psoriasis within 30 days of Visit 1.
5. Subject has used any of the following systemic medications or procedures:

   * Systemic tofacitinib, ampremilast, methotrexate, retinoids, corticosteroids, and cyclosporine or analogous products with in three months of Visit I; or
   * Systemic anti-inflammatory biologic therapy (i.e., FDA-approved or experimental therapy) with in five half-lives of the biologic prior to Visit 1.
6. Subject is currently using lithium or Plaquenil.
7. Subject is currently using a beta-blocking medication (e.g., propranolol) or angiotensin converting enzyme (ACE) inhibitor at a dose that has not been stabilized, in the opinion of the investigator.
8. Subject, in the opinion of the investigator, has had prolonged exposure to natural or artificial sources of ultraviolet (UV) radiation within 30 days prior to Visit 1 or intends to have such exposure during the study that is likely to modify the subject's disease.
9. Subject is currently enrolled in an investigational drug or device study.
10. Subject has used an investigational drug or investigational device treatment within 30 days prior to first application of the test article.
11. Subject has a history of sensitivity to any of the ingredients in the test article.
12. Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2018-02-13 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in sum of clinical signs of psoriasis (scaling, erythema, and plaque elevation) scores. | Day 29
  Scaling, erythema and plaque elevation will each be scored on a 5-point scale where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe. These evaluations are an assessment of the overall or "average" degree of each of three key characteristics present within all of the subject's psoriatic lesions in the Treatment Area by the investigator or designee.

SECONDARY OUTCOMES:
The proportion of subjects with improvement versus Baseline in IGA score. | Day 29
  The Investigator's Global Assessment (IGA) will be assessed on a 5-point scale where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe.
The proportion of subjects with improvement versus Baseline for each of the clinical signs of psoriasis (scaling, erythema and plaque elevation) | Day 29

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Site 03, Tampa, Florida
  - Site 04, Carmel, Indiana
  - Site 05, Plainfield, Indiana
  - Site 02, Albuquerque, New Mexico
  - Site 01, High Point, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided